CLINICAL TRIAL: NCT06354790
Title: A Prospective, Longitudinal, Interventional Natural History Study of Children With LAMA2-related Dystrophies
Brief Title: Natural History Study of Children With LAMA2-related Dystrophies
Acronym: LAMA2
Status: Recruiting | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NatHis LAMA2
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Merosin Deficient Congenital Muscular Dystrophy
Keywords: LAMA2; Congenital Muscular Dystrophy; Natural history
MeSH Terms: conditions — Muscular dystrophy congenital, merosin negative | interventions — Mental Status and Dementia Tests; Respiratory Physiological Phenomena; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Other: Motor evaluations; Other: Cognitive assessment; Other: Pulmonary function test; Other: Cardiac evaluation; Other: Quality of life; Other: Spine X Ray; Other: Muscular MRI; Other: Biomarkers collection and analysis

INTERVENTIONS:
Other: Motor evaluations — Evaluation of patients motor function using motor scales (MFM32, RULM), Timed functioned tests (6MWT, Rise from floor, 4SCT, 10mWT), dynamometric strength evaluation (grip, pinch, flexion/extension)
Other: Cognitive assessment — Patients cognitive evaluation (WPPSI-IV, WISC-V)
Other: Pulmonary function test — Evaluation of patients' respiratory function (FVC, PCF, MIP, MEP, SNIP)
Other: Cardiac evaluation — Evaluation of patients' cardiac function (ECG, Echo-cardiography)
Other: Quality of life — Evaluation of patients quality of life with questionnaires and PROM
Other: Spine X Ray — Evaluation of spinal deformities by X-ray
Other: Muscular MRI — Evaluation of a qualitative whole-body muscle part and a quantitative lower limb muscle part by MRI
Other: Biomarkers collection and analysis — Collection of blood and urinary sample for biomarkers research.

SUMMARY:
The goal of this natural history study is to characterize the disease course, characteristics in paediatric population of LAMA2-RD (related dystrophies) patients.

The aim of the study is to establish a well-described cohort of patients in France with LAMA2-RD for prospective follow-up and recruitment for future clinical trials.

Participants will be follow up during a two years period regarding exhaustive aspects of the pathology:

* Muscular function
* Respiratory function
* Cognitive phenotyping
* Quality of life
* Growth parameters
* Biomarkers

DETAILED DESCRIPTION:
The international workshop on LAMA2-RD, held in 2019 in Maastricht, stressed the importance of the identification of LAMA2-RD patients and the natural history studies worldwide. Together with the recent progress in preclinical applications, the road to therapy is paved.

However, no effective treatment has currently received market approval. Given the phenotype variability in LAMA2-RD patients, even in very young ones, determining which outcome measure(s) could be the most appropriate to assess the efficacy of potential therapies, and which variables are prognostic of the disease course, is required. In consequence, it is clearly necessary to explore all the aspects of the pathology: physiological, clinical/motor, biological, aligning with current or future international studies though collaboration.

Unlike results obtained through a retrospective study, data from a prospective natural history will be less subject to bias and error. Control of the studied population will also lead to reduce the variability of the results. The different variables explored during this study aim to cover all aspects of the disease and appear to be relevant candidates as outcomes.

The aim of the study is to focus on the clinical phenotyping and to establish a well-described cohort of patients in France with LAMA2-RD for prospective follow-up and recruitment for future clinical trials. One other objective is to validate the use of a large subset of outcome measures in LAMA2-RD. Adding an electrophysiological data will give more insight to the neuropathology of the disease and enlarge the scope of futures therapies.

An exploratory part will test if denaturation profiling of plasma from patients can be used to follow disease progression. Finally, serum and plasma samples from patients will also be stored for future studies focused on searching and validating novel biomarkers in LAMA2-RD.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the Legal Authority Responsible and/or assent by the subject (starting from 6 years old)
* Subject must be
* Supportive clinical phenotype and diagnosis of LAMA2-RD, confirmed by:

  * Two pathogenic variants in the LAMA2 gene (via a diagnostic laboratory included on an approved list of genetic testing laboratories (Annex 1)) or
  * Muscle biopsy with absence of merosin (laminin-211) and at least one pathogenic variant in the LAMA2 gene
* Absence of another confirmed neurological genetic disease
* Willingness to maintain current exercise and/or physical therapy regimen for the duration of the clinical study
* Willingness to comply with the study protocol, including all the mandatory study procedures and visits
* Affiliated to or a beneficiary of a French or acknowledged in France, social security scheme

Exclusion Criteria:

* Developmental quotient less than 70 and/or behavioral disorder requiring general anesthesia to perform an MRI
* Acute medical illness or hospitalization within 30 days prior to informed consent
* Participation in a previous trial of any investigational agent for LAMA2-RD, or use of any other investigational therapy within 30 days prior to informed consent, or participation in other clinical studies, within 30 days (or 5 half-lives, whichever is longer) prior to informed consent, which, in the opinion of the PI, may potentially confound results from this study
* Other significant medical condition and/or overall fragility of medical status, which in the opinion of the Investigator may confound interpretation of the clinical course of LAMA2-RD
* Pregnant or breastfeeding women

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 young patients aged between 2 and 15 years old (inclusive) at time of consent, with a confirmed LAMA2 diagnosis (muscle biopsy with absence of merosin (laminin-211) and at least one pathogenic variant in the LAMA2 gene)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-12-04 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Motor function Measurement (MFM32) score | Through study completion, an average of 2 years
Change in Motor Milestone Checklist | Through study completion, an average of 2 years
  Acquisitions and losses of motor functions (ex: Head control, sitting, crawling, standing, walking, climbing stairs, jumping,running, hopping,...)
Change in Revised Upper Limb Module (RULM) score | Through study completion, an average of 2 years
Change in grip strength measured by dynamometer tool | Through study completion, an average of 2 years
Change in pinch strength measured by dynamometer tool | Through study completion, an average of 2 years
Change in arm flexion/extension strength measured by dynamometer tool | Through study completion, an average of 2 years
Change in 6 Minutes Walking Test | Through study completion, an average of 2 years
Change in 4 Stairs Climbing Test (4SCT) | Through study completion, an average of 2 years
Change in 10m Walking Test | Through study completion, an average of 2 years
Change in Rise from Floor Test | Through study completion, an average of 2 years
Change in patient's Forced Vital Capacity (FVC) results | Through study completion, an average of 2 years
Change in patient's Peak Cough Flow (PCF) results | Through study completion, an average of 2 years
Change in patient's Maximum Expiratory Pressure (MEP) results | Through study completion, an average of 2 years
Change in patient's Maximal Inspiratory Pressure (MIP) results | Through study completion, an average of 2 years
Change in patient's Sniff Nasal Inspiratory Pressure (SNIP) results | Through study completion, an average of 2 years
Change in patient's muscle fat replacement measured by Magnetic Nuclear Resonance | Through study completion, an average of 2 years
Change in patient's cross-sectional area of the residual muscle measured by MNR | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Change in Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV) results | Through study completion, an average of 2 years
Change in Wechsler Intelligence Scale for Children-V (WISC-V) results | Through study completion, an average of 2 years
Change in PedsQL questionnaire results | Through study completion, an average of 2 years
Change in CGI-S questionnaire results | Through study completion, an average of 2 years
Change in CGI-I questionnaire results | Through study completion, an average of 2 years
Change in Faces pain rating scale results | Through study completion, an average of 2 years
Change in Fatigue Severity Scale results | Through study completion, an average of 2 years
Change in ACTIVLIM questionnaire results | Through study completion, an average of 2 years
Change in Egen Klassifikation Scale Version 2 (EK2) results | Through study completion, an average of 2 years
Change in Caregiver burden questionnaire (LMDIS) results | Through study completion, an average of 2 years
  LAMA2 Dystrophy Independence Scale

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre de Référence GNMH, Pédiatrie Hôpital Raymond-Poincaré, Garches
  - Service de MPR pédiatrique L'Escale - HCL, Lyon
  - Département de neuropédiatrie Pôle Femme Mère Enfant CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Plateforme d'essais cliniques pédiatriques iMotion, Paris

IPD SHARING:
Plan to Share IPD: No